CLINICAL TRIAL: NCT04353570
Title: Psychological Impact of Confinement on the Adult Population Followed in Outpatient Psychiatry at EPS Ville Evrard: Three-month Longitudinal Clinical Evaluation
Brief Title: Psychological Impact of Confinement on the Adult
Acronym: IMPA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre hospitalier de Ville-Evrard, France (Other)
Responsible Party: Principal Investigator, Januel, clinical research unit director, Centre hospitalier de Ville-Evrard, France
Other Study IDs: 10477M-IMPA
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Identify the Psychological Impact of Containment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: clinical interview — This interview can be carried out face to face or remotely. In the latter case, it is part of telemedicine, which is recognised by the health authorities in France.

SUMMARY:
This clinical interview is made to allow a clinical follow-up of the patients followed in psychiatry of the EPS Ville-Evrard establishment in a simple way and in a secure medical framework during the period of the epidemic and the confinement from March 30 to June 30, 2020.

ELIGIBILITY:
Inclusion Criteria:

Adult patient followed in outpatient psychiatry at EPS Ville Evrard and agrees to participate -

Exclusion Criteria:

Adult patient followed in outpatient psychiatry at EPS Ville Evrard and does not wish to participate

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patient followed in outpatient psychiatry at EPS Ville Evrard
Sampling Method: Non-Probability Sample
Enrollment: 2100 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-06-18 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Depression MINI DIAG and Anxiety questionnaire and the The Global Performance Rating Scale and CGI-truth | three month

CONTACTS AND LOCATIONS:
Locations (1):
- Unité de recherche clinique, Neuilly-sur-Marne, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No